CLINICAL TRIAL: NCT03088683
Title: Comparison of Liver Trauma in Two Retractors Used in Sleeve Gastrectomy: A Prospective Multicenter Clinical Trial
Brief Title: Comparison of Liver Trauma in Two Retractors Used in Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah Sisik, General Surgery Specialist, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMP-LIV-RET
Record Dates: First submitted 2017-01-16; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: sleeve gastrectomy; liver retractor; nathanson; reveel; liver trauma
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nathanson Retractor (Active Comparator): Nathanson retractor will be used
  Interventions: Device: Nathanson Retractor
- Reveel Retractor (Active Comparator): Reveel retractor will be used
  Interventions: Device: Reveel Retractor

INTERVENTIONS:
Device: Nathanson Retractor — Liver will be retracted with Nathanson retractor
  Arms: Nathanson Retractor
Device: Reveel Retractor — Liver will be retracted with Reveel retractor
  Arms: Reveel Retractor

SUMMARY:
In Laparoscopic Sleeve Gastrectomy, retraction of the left lobe of the liver is important for an effective visualisation. There are many retractors available for this retraction. A study is designed to compare two different liver retractors for liver trauma; Nathanson liver retractor that is used more commonly and Reveel liver retractor that has more recent history of use.

DETAILED DESCRIPTION:
A randomised controlled prospective study is designed with 80 patients over 3-month period (January 2017 to March 2017). Laparoscopic sleeve gastrectomy is planned for all patients. Two groups are designed depending on retractor. Liver retraction will be provided with Nathanson retractor in first group (Nathanson group, 40 patients), and with Reveel retractor in second group (Reveel group, 40 patients). Preoperative serum levels of transaminases, total bilirubin and C-reactive protein will be measured in all patients. The same biochemical markers will be measured on days 1 and 2 postoperatively. The patients with body mass index (BMI) ≥35kg/m2 are enrolled to study. The parameters of demographic characteristics (age, gender, BMI, weight, and body fat percentage), and clinical outcomes (postoperative complications, mortality, readmissions) are planned to record.

Operative Technique

All patients will be operated by same surgeons. and anesthetist. Peroperatively intravenous paracetamol 10 mg, tramadol 50 mg and fentanyl 150 mcg will be used for analgesia. Laparoscopic sleeve gastrectomy will be performed with 5 trocars, in reverse trendelenburg position by creating pneumoperitoneum with 14 mmHg carbon dioxide insufflation. Trocar replacements are one 10-mm trocar in the midline above umbilicus for the endoscope, one 12-mm trocar to right midclavicular line linage to the 10-mm trocar. One 5-mm trocar to the left midclavicular line linage to the 10-mm trocar, one 5-mm trocar to the front axillary line below the left costal margin. Both liver retractors will be placed from 2 cm below the xiphoid process for liver retractor. In nathanson group; after placing the blade of Nathanson retractor below the left lobe of the liver, it will be fixed to the operating table by the other instruments of retractor. In reveel group; the retractor will be placed below the left lobe of the liver and then it will be fixed to the skin with a towel clamp. 38 F orogastric tube will be used. No use of nasogastric tubes and urinary catheters routinely is planned. Drain replacement is planned for all patients.

Preoperative and postoperative values of the markers will be analysed and compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with BMI>35

Exclusion Criteria:

* patients with known liver disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04-01 (Estimated); Study Completion 2017-04-20 (Estimated)

PRIMARY OUTCOMES:
Changes in physiological parameters of liver due to trauma of retractors | within the first 2 days of the surgery
  Traumatic effects of liver retractors in sleeve gastrectomy. Number of participants with abnormal laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Sisik, Principal Investigator — Umraniye Education and Research Hospital
Locations (1):
- Nazif Bagriacik Kadioy Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided